CLINICAL TRIAL: NCT07235514
Title: General Anesthesia Versus Procedural Sedation in Endovascular Therapy for Anterior Circulation Large Vessel Occlusion Stroke: A Multicenter Prospective Randomized Trial
Brief Title: Anesthesia Management in Endovascular Therapy for Ischemic Stroke - 2
Acronym: AMETIS 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: PHRC, Ministry of Health France (Unknown); STROKELINK (Unknown); ANARLF Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC 2024 CHABANNE; 2025-A00169-40 (Other: 2025-A00169-40)
Record Dates: First submitted 2025-10-02; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke; Anterior Cerebral Circulation; General Anesthesia; Procedural Sedation; Thrombectomy
Keywords: Ischemic stroke; anterior circulation; mechanical thrombectomy; anesthetic strategy; general anesthesia; procedural sedation; functional outcome; large vessel occlusion stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open Blinded Endpoint trial (PROBE design)
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Experimental): General anesthesia with intubation and mechanical ventilation:
  ECG, SpO2 and BP. BP will be measured every 2 minutes Hyperglycemia (>180mg/dL) and hypoglycemia (<60mg/dL) should be treated (outside of the protocol)
  Systolic BP: 150 - 180mmHg with Diastolic BP < 105mmHg Norepinephrine tartrate infusion or Nicardipine on a peripheral intravenous line or on a 3-way venous extender, as necessary EtCO2 35 - 45mmHg SpO2 above 94 %. Glycemia as needed
  End of procedure: Anesthesia will be immediately stopped and extubation should not be delayed. After the intervention, patients are transferred to the post anesthesia care unit and are then admitted to the stroke unit
  First 24 hours: SBP<180mmHg, DBP<110mmHg and MAP>65mmHg, SpO2 > 94 %, temperature < 38°C, blood glucose 60 - 180mg/dL. Other aspects of monitoring are not modified by the protocol.
  24-48h outside of the protocol: non-contrast brain CT or a brain MRI
  Interventions: Procedure: General Anesthesia
- Procedural sedation (Experimental): Procedural sedation with spontaneous ventilation:
  ECG, SpO2 and BP. BP will be measured every 2 minutes Hyperglycemia (>180mg/dL) and hypoglycemia (<60mg/dL) should be treated (outside of the protocol)
  Systolic BP: 150 - 180mmHg with Diastolic BP < 105mmHg Norepinephrine tartrate infusion or Nicardipine on a peripheral intravenous line or on a 3-way venous extender, as necessary Breathing face mask: EtCO2 and oxygen as necessary SpO2 above 94 %. Glycemia as needed
  End of procedure: Procedural sedation will be immediately stopped. After the intervention, patients are transferred to the post anesthesia care unit and are then admitted to the stroke unit
  First 24 hours: SBP<180mmHg, DBP<110mmHg and MAP>65mmHg, SpO2 > 94 %, temperature < 38°C, blood glucose 60 - 180mg/dL. Other aspects of monitoring are not modified by the protocol.
  24-48h outside of the protocol: non-contrast brain CT or a brain MRI
  Interventions: Procedure: Procedural sedation

INTERVENTIONS:
Procedure: General Anesthesia — In the general anesthesia (GA) group with tracheal intubation : Clinical target: unarousable state Standard preoxygenation, • Rapid sequence induction of GA will use intravenous Etomidate (0.2-0.3mg/Kg) or Ketamine (1-2mg/Kg) and Succinylcholine (1mg/Kg) or Rocuronium (1.2 mg/Kg) • Maintenance of GA will use intravenous Propofol (brain tissue target controlled infusion up to 4.0 µg/mL or up to 5.0 mg/kg/hr) or Sevoflurane (end-tidal concentration up to 2% (EtSevo)) and intravenous Remifentanil (brain tissue target controlled infusion up to 4.0 ng/mL) Movement despite unarousable state: NMBA as needed
  Other Names: GA
  Arms: General anesthesia
Procedure: Procedural sedation — In the procedural sedation group with spontaneous ventilation :
  Clinical target: alert and "confortable" i.e. minimal to moderate sedation level
  * Subcutaneous local anesthesia with Lidocaine 10mg/mL (maximum 10mL)
  * Intravenous Remifentanil as necessary to achieve the sedation clinical target (brain tissue target controlled infusion up to 2.0 ng/mL). Propofol could be added as necessary (brain tissue target controlled infusion up to 3.0 µg/mL or 2.0 mg/kg/hr).
  The lightest sedation level allowing the intervention has to be sought.
  Other Names: PS
  Arms: Procedural sedation

SUMMARY:
The goal of this clinical trial is to learn what is the best anesthetic management in participants with severe stroke that require a medical intervention called mechanical thrombectomy (MT) done to open the occluded brain vessel.

The main question it aims to answer is:

• Is general anesthesia (GA) better than procedural sedation (PS) for improving functional performance and decrease dependance in daily life 3 months after stroke?

GA (a non-arousable state induced by anesthetic medications that require respiratory assistance) or PS (a state of reduced arousal induced by lesser dose of anesthetic medications that do not require respiratory assistance) are both used for MT. GA enables strict immobility that could facilitate the conduct of MT but lessen blood pressure and blood flow in the brain. PS provides less drop in blood pressure but MT could be more difficult due to possible movement and breathing may be decreased.

Researchers will compare GA with PS to see which one is better for MT success and for the functional consequences of stroke.

Participants will be treated with GA or PS for the intervention of MT and will be followed by researchers during their hospital stay and asked by a telephone interview how is their functional status 3 months after stroke.

DETAILED DESCRIPTION:
Mechanical thrombectomy (MT) has significantly improved the outcome of anterior circulation large vessel occlusion stroke. The MT procedure could require management by a dedicated anesthesia team to ensure safety and immobility of these frail patients, in order to quickly restore cerebral perfusion and prevent procedural complications. The anesthetic strategy (general anesthesia with tracheal intubation (GA) or procedural sedation with spontaneous ventilation (PS)) can impact the conduct of the procedure and influence the functional outcome. GA ensures immobility and airway control, but can alter blood pressure (BP). PS provides better control of BP but may be associated with respiratory failure and movements that could interfere with intra-arterial navigation.

Three European single-center randomized controlled trials (RCTs) found no difference between GA and PS for their respective primary endpoints. These three trials were pooled in an individual patient data meta-analysis that evaluated functional outcome (modified Rankin Scale mRS) at 3 months as the primary endpoint. 368 patients were included, and GA was associated with a better functional outcome (mean mRS score was 2.8 (95% CI, 2.5-3.1) in the GA group vs. 3.2 (95% CI, 3.0-3.5) in the PS group (difference, 0.43 [95% CI, 0.03-0.83])). The main limitations of this trial were 1) the small sample size (3 small single-center trials), 2/ a possible center effect with over-representation of one trial on the primary endpoint, and 3/ a highly selected population (exclusion of less severe patients (NIHSS<10), stroke presentation > 8 hours and wake up stroke).

Two French multicenter RCTs have recently been published. The GASS trial included 345 patients in four centers with dedicated GA and PS protocols. There was no difference in the primary endpoint, which was functional independence (mRS 0 to 2) at three months (36% for PS vs. 38% for GA (RR, 0.91 [95% CI, 0.69 to 1.19], p = 0.47)). The AMETIS trial included 273 patients in 10 centers with no specified GA or PS protocol. There was no difference in the primary endpoint, which was a composite of functional independence at 3 months and absence of any peri-procedural and medical complications during the first 7 days. The median mRS was 3 (2-5) under GA vs. 3 (2-4) under PS; RR 0.80 [95% CI: 0.53 to 1.22]. GA was strongly associated with the occurrence of arterial hypotension (87.4% vs. 44.9% in the PS group).

However, 1) these multicenter trials had relatively small sample sizes, 2) the time of assessment of the primary outcome measure was highly variable in GASS, and 3) in AMETIS, the BP targets in the GA group were not met and there was heterogeneity in drug management under PS and GA.

These contradictory results reveal a persistent clinical equipoise regarding this important issue.

The AMETIS-2 trial will evaluate almost every patient with anterior circulation large vessel occlusion stroke eligible for MT in different French comprehensive stroke centers.

The trial protocol for PS and GA will use dedicated anesthetic and hemodynamic management protocols.

The primary outcome measure will use an ordinal shift analysis of the mRS score evaluated at 3 months as the primary endpoint.

To extend the effect analysis, functional independence, cognitive and quality of life assessment will be evaluated as secondary endpoints at 3 months.

We therefore hypothesize that, with a dedicated anesthetic protocol and strict hemodynamic control, GA will lead to a better long-term functional outcome after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute ischemic stroke with an occlusion of the intracranial internal carotid artery and/or the proximal middle cerebral artery (M1-M2) with or without association of extracranial occlusion of the cervical internal carotid artery (tandem lesion)
* Eligible for mechanical thrombectomy according to international guidelines
* Informed and signed consent of patient, or if he is unable to consent the consent of patient's relative or emergency procedure in the absence of relative
* National health insurance

Exclusion Criteria:

* Coma or altered vigilance defined as a score ≥ 2 on the level of consciousness 1A subscale of the NIHSS
* Premorbid disability defined as a mRS > 2
* Posterior circulation stroke
* Associated cerebral hemorrhage
* Stroke complicating another acute illness or postoperative stroke
* Emesis at arrival in angiosuite
* Allergy to anesthetic medication
* Pregnant or breast-feeding women
* Adult under the protection of the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | Day 90 after the stroke
  modified Rankin Scale, that range from 0 to 6: 0, no neurologic deficit; 1, no clinically significant disability; 2, slight disability; 3, moderate disability requiring some help; 4, moderately severe disability; 5, severe disability; 6, death
  > measured centrally by a blinded evaluator

SECONDARY OUTCOMES:
Functional independence = key secondary outcome | Day 90 after the stroke
  Functional independence defined as a score of 0-2 on the rating of the modified Rankin Scale measured centrally by a blinded evaluator. This will be analyzed as a dichotomized measure
Modified Treatment in Cerebral Infarction scale at the end of thrombectomy (mTICI). | At day 1 (end of the thrombectomy procedure)
  To assessed efficacy of GA vs PS
Good quality of reperfusion defined as a mTICI score of 2b-3 | At day 1 (end of the thrombectomy procedure)
  To assessed efficacy of GA vs PS
Excellent quality of reperfusion defined as a mTICI score of 2c-3 | At day 1 (end of the thrombectomy procedure)
  To assessed efficacy of GA vs PS
National Institute of Health Stroke Scale (NIHSS) | At day 1 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
National Institute of Health Stroke Scale (NIHSS) | At day 7 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Length of stay in stroke-unit and hospital | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
moderate recovery defined as a score of 0-3 on the rating of the modified Rankin Scale | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Utility-weighted modified Rankin scale | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Barthel index | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Montreal Cognitive Assessment (MOCA) | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Stroke Specific Quality Of Life scale (SSQOL) | At day 90 after the thrombectomy procedure
  To assessed efficacy of GA vs PS
Per-interventional arterial dissection or perforation defined as a flow-limiting tear or flap in the arterial wall or arterial extravasation of contrast media | At the end of the thrombectomy procedure
  To assessed safety of GA vs PS
Per-interventional embolization in another territory defined as a new (not present on the first angiogram) arterial occlusion outside of the middle cerebral artery territory | At the end of the thrombectomy procedure
  To assessed safety of GA vs PS
Procedural hypotension, hypertension, blood pressure variability, hypoxemia and aspiration (Yes or No) | At the end of the thrombectomy procedure
  To assessed safety of GA vs PS
Hemodynamic protocol adherence | At day 1 after the thrombectomy procedure
  To assessed safety of GA vs PS
Post-interventional groin hematoma defined as an accumulation of blood at the puncture site requiring evacuation, transfusion, or extended hospital stay | At day 7 after the thrombectomy procedure
  To assessed safety of GA vs PS
Intracranial hemorrhage | At day 1 after the thrombectomy procedure
  To assessed safety of GA vs PS
medical complications (could be evaluated before day 7 if the patient quit the hospital) | At day 7 after the thrombectomy procedure
  To assessed safety of GA vs PS
Mortality | At day 7 after the thrombectomy procedure
  To assessed safety of GA vs PS
Mortality | At day 90 after the thrombectomy procedure
  To assessed safety of GA vs PS

CONTACTS AND LOCATIONS:
Overall Officials: Russell CHABANNE, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication can be made available upon specific request from investigators.

REFERENCES:
- [Background] Schonenberger S, Henden PL, Simonsen CZ, Uhlmann L, Klose C, Pfaff JAR, Yoo AJ, Sorensen LH, Ringleb PA, Wick W, Kieser M, Mohlenbruch MA, Rasmussen M, Rentzos A, Bosel J. Association of General Anesthesia vs Procedural Sedation With Functional Outcome Among Patients With Acute Ischemic Stroke Undergoing Thrombectomy: A Systematic Review and Meta-analysis. JAMA. 2019 Oct 1;322(13):1283-1293. doi: 10.1001/jama.2019.11455. PMID 31573636
- [Background] Chabanne R, Geeraerts T, Begard M, Balanca B, Rapido F, Degos V, Tavernier B, Molliex S, Velly L, Verdonk F, Lukaszewicz AC, Perrigault PF, Albucher JF, Cognard C, Guyot A, Fernandez C, Masgrau A, Moreno R, Ferrier A, Jaber S, Bazin JE, Pereira B, Futier E; ANARLF NetworkAMETIS Study Group. Outcomes After Endovascular Therapy With Procedural Sedation vs General Anesthesia in Patients With Acute Ischemic Stroke: The AMETIS Randomized Clinical Trial. JAMA Neurol. 2023 May 1;80(5):474-483. doi: 10.1001/jamaneurol.2023.0413. PMID 37010829
- [Background] Maurice A, Eugene F, Ronziere T, Devys JM, Taylor G, Subileau A, Huet O, Gherbi H, Laffon M, Esvan M, Laviolle B, Beloeil H; GASS (General Anesthesia versus Sedation for Acute Stroke Treatment) Study Group and the French Society of Anesthesiologists (SFAR) Research Network. General Anesthesia versus Sedation, Both with Hemodynamic Control, during Intraarterial Treatment for Stroke: The GASS Randomized Trial. Anesthesiology. 2022 Apr 1;136(4):567-576. doi: 10.1097/ALN.0000000000004142. PMID 35226737
- [Background] Quintard H, Degos V, Mazighi M, Berge J, Boussemart P, Chabanne R, Figueiredo S, Geeraerts T, Launey Y, Meuret L, Olivot JM, Pottecher J, Rapido F, Richard S, Saleme S, Siguret-Depasse V, Naggara O, De Courson H, Garnier M. Anaesthetic and peri-operative management for thrombectomy procedures in stroke patients. Anaesth Crit Care Pain Med. 2023 Feb;42(1):101188. doi: 10.1016/j.accpm.2022.101188. Epub 2023 Jan 1. PMID 36599377
- [Background] Turc G, Bhogal P, Fischer U, Khatri P, Lobotesis K, Mazighi M, Schellinger PD, Toni D, de Vries J, White P, Fiehler J. European Stroke Organisation (ESO) - European Society for Minimally Invasive Neurological Therapy (ESMINT) Guidelines on Mechanical Thrombectomy in Acute Ischaemic StrokeEndorsed by Stroke Alliance for Europe (SAFE). Eur Stroke J. 2019 Mar;4(1):6-12. doi: 10.1177/2396987319832140. Epub 2019 Feb 26. PMID 31165090
- [Background] Powers WJ, Rabinstein AA. Response by Powers and Rabinstein to Letter Regarding Article, "2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association". Stroke. 2019 Sep;50(9):e277-e278. doi: 10.1161/STROKEAHA.119.026917. Epub 2019 Aug 8. No abstract available. PMID 31390963